CLINICAL TRIAL: NCT02385565
Title: Effect Of The System In The Enriched Fat Metabolism Of The Child Reached Mitochondrial Cytopathy
Acronym: MITOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2004/0401; 2004/0138 (Other: DGS)
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Mitochondrial Cytopathies Disorders
MeSH Terms: interventions — Diet, High-Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- high fat diet (Experimental): 10 % proteins, 30 % lipids, 60 % carbohydrates
  Interventions: Other: high fat diet
- Normal fat diet (Placebo Comparator): 10 % proteins, 45 % lipids, 45 % carbohydrates
  Interventions: Other: normal fat diet

INTERVENTIONS:
Other: high fat diet — high fat diet as 10 % proteins, 30 % lipids, 60 % carbohydrates
  Arms: high fat diet
Other: normal fat diet — high fat diet as 10 % proteins, 45 % lipids,45 % carbohydrates
  Arms: Normal fat diet

SUMMARY:
The aim of the present study is to compare Resting Energy Expenditure (REE) between normal fat diet (NFD) as a control vs high fat diet (HFD) as a treatment in Mitochondrial cytopathies disorders ( MID's ) patients. Secondary objectives is to compare diet induced thermogenesis (DIT) and body composition between NFD vs HFD.

This study is a randomized cross-over study. Normal fat diet (ie 10 % proteins, 45 % lipids, 45 % carbohydrates) is the imposed diet at baseline, high fat diet (ie 10 % proteins, 30 % lipids, 60 % carbohydrates is used according to the cross-over design trial. Main evaluation criteria is REE and second evaluation criteria is DIT both measured by indirect calorimetry ). 36 included MID subjects will be included in this study. Main evaluation criteria and second evaluation criteria will be measured at baseline, 1 month, 2 month and 3 month.

DETAILED DESCRIPTION:
REE and DIT are measured by indirect calorimetry . The device used is a using an open-circuit ventilated hood system (QUARK RMR®, Cosmed, Pavona; Italy). The respiration quo- tient (RQ) and flow settings are calibrated by reference to alcohol combustion every six months. Before each test, the calorimeter is calibrated with a reference gas mixture (5% CO2, 95% O2 v/v). Expired carbon di- oxide (VCO2) and inspired oxygen (VO2) -flows are recorded, as well as the RQ. EE is calculated every minute from oxygen consumption (VO2 in ml/min) and carbon dioxide production (VCO2 in ml/min) using the Weir formula without protein correction. DIT is measured during 6 hours after a calibrated breakfast (normal fat diet or high fat diet according to the cross-over design) as 30% of theoric energy intake.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 21 years-old children,

  * Children with a proven mitochondrial cytopathy documented on biopsies by histology, histoenzymology, ultrastructure and enzyme assay and/or on body fluids by laboratory markers including lactacidemia, metabolic acidosis, increased CSF lactate, lactate/pyruvate and beta-hydroxybutyrate/acetoacetate ratios, paradoxical postprandial ketonemia, alaninemia, citrullinemia, plasma acylcarnitines.
  * Children on the usual diet (30% lipids, 60% glucides and 10% proteins) for at least 1 month.
  * Informed consent of the 2 parents and from the child when in age to express a consent.
  * Child with a social security cover.

Exclusion Criteria:

* Acute infection (fever > 38.5°C for more than 6h) within 7 days prior to the study.
* Disability for understanding and following the protocol
* Rejection of the study by the patient or failure to comply to the protocol

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2004-02; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
resting energy expenditure | up to 3 months
  resting energy expenditure measured by indirect calorimetry

SECONDARY OUTCOMES:
diet induced thermogenesis | baseline, 1 month, 2 months, 3 months
  diet induced thermogenesis measured by indirect calorimetry
body composition | baseline, 1 month, 2 months, 3 months
  body composition by DEXA

CONTACTS AND LOCATIONS:
Overall Officials: Dries DOBBELAERE, MD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Centre d'Investigation Clinique, Lille
  - Centre d'Investigation Clinique, Paris